CLINICAL TRIAL: NCT01881048
Title: Window of Opportunity Study Targeting the Inflammatory Milieu of Pregnancy Associated Breast Cancer
Brief Title: Window of Opportunity Study Targeting the Inflammatory Milieu
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-0104.cc; NCI-2011-02967 (Other: National Cancer Institute)
Record Dates: First submitted 2013-06-14; First posted 2013-06-19 (Estimated); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Stage IA Breast Cancer; Stage IB Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer
Keywords: Breast cancer; Omega-3 Fatty Acid; Celecoxib; Celebrex; Surgery
MeSH Terms: conditions — Breast Neoplasms | interventions — Fatty Acids, Omega-3; Fish Oils; Docosahexaenoic Acids; Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (No Intervention): Patients undergo observation.
- Arm II (fish oil) (Experimental): Patients receive omega-3 fatty acid by mouth everyday until the morning of surgery.
  Interventions: Dietary Supplement: Omega-3 fatty acid
- Arm III (celecoxib) (Experimental): Patients receive celecoxib by mouth twice a day until the morning of surgery.
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Dietary Supplement: Omega-3 fatty acid — Given PO
  Other Names: fish oil, n-3 fatty acid, omega-3 polyunsaturated fatty acid
  Arms: Arm II (fish oil)
Drug: Celecoxib — Given PO
  Other Names: Celebrex
  Arms: Arm III (celecoxib)

SUMMARY:
The purpose of this study is to evaluate the effect of two anti-inflammatory drugs, fish oil capsules and the COX-2 inhibitor celecoxib, on pregnancy associated breast cancer (PABC). Short-term intervention with anti-inflammatory medications will demonstrate a reduction in the inflammation and immune suppressive phenotype of PABC, and decreased metastatic potential in PABC. This unique window in breast cancer management serves as a valuable opportunity to obtain preliminary data on biomarkers and the alterations that occur when the system is troubled by a drug or other intervention which will be instrumental in designing future therapeutic or preventative strategies for larger clinical study.

DETAILED DESCRIPTION:
This randomized pilot clinical trial studies omega-3 fatty acid or celecoxib in treating patients with breast cancer planning to undergo surgery. Omega-3 fatty acid may stimulate the immune system in different ways and stop tumor cells from growing. Celecoxib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether omega-3 fatty acid or celecoxib is more effective in treating breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age greater or equal to 18 and less than or equal to 50.
* Histological or cytological confirmation of breast cancer; for patients with fine needle aspiration (FNA), a core biopsy must be intended
* For patients diagnosed with needle core or excisional biopsy, formalin-fixed paraffin embedded tumor blocks or unstained slides must be available or patient must be willing to undergo repeat core biopsy for research purposes as part of study procedures (biopsy for fresh/ fresh frozen tissue is otherwise optional)
* Any clinical stage allowed provided definitive local resection intended and neoadjuvant treatment not intended
* Patient must be planned to proceed to definitive surgery for their breast cancer at least 1 week or more after diagnosis
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Patient must have laboratory parameters as follows:
* Liver function tests (Total bilirubin, aspartate aminotransferase, alanine aminotrasferase, alkaline phasphataseAST) =< 2 x ULN
* Platelet count greater than or equal to institutional lower limit of normal (LLN)
* Patient cannot have greater than grade 1 anemia as determined by hematocrit (Hct)
* Written informed consent obtained prior to any initiation of study procedures
* Willingness to abstain from either fish oil or celebrex for study period if randomized to control arm
* Women who are lactating at time of diagnosis are eligible provided they complete weaning prior to starting study drug

Exclusion Criteria:

* Known autoimmune condition, chronic steroid use, underlying immune disease (other than breast cancer), use of immunomodulatory prescription drugs for any medical condition
* Known allergy or intolerance to fish oil, fish, non-steroidal anti-inflammatory drugs (NSAIDS), acetylsalicylic acid (ASA) or cyclooxygenase-2 (COX 2) inhibitors
* Known bleeding diathesis or history of peptic ulcer disease; gastroesophageal reflux allowed if controlled
* Currently taking greater than one 1000mg fish oil capsule daily or celecoxib at baseline, unless willing to stop consumption 1 week prior to starting study
* History of stroke, transient ischemic attack (TIA) or coronary artery disease
* The presence of other comorbid conditions known to impact immune function, (such as: type I diabetes, uncontrolled adult onset diabetes, severe chronic obstructive pulmonary disease (COPD), uncontrolled infection or known human immunodeficiency virus [HIV] infection)
* Underlying psychiatric condition which would, in the opinion of the investigator, preclude compliance with study requirements
* Women who are pregnant at time of breast cancer diagnosis and intend to continue the pregnancy; if pregnancy is terminated per patient's cancer decision making, they would be eligible for participation afterwards
* History of other malignancy besides current diagnosis of breast cancer, unless definitively treated more than 5 years ago
* Any history of Hodgkin's disease requiring mantle field irradiation
* Any previous diagnosis of breast cancer

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 42 (Actual)
Dates: Start 2009-12-08 (Actual); Primary Completion 2014-01-14 (Actual); Study Completion 2015-12-14 (Actual)

PRIMARY OUTCOMES:
Change in mean Ki-67 index in patients receiving either omega-3 fatty acid or celecoxib for 1 or more weeks as compared to controls | Baseline and 1 week
  Tumor cells are stained using the Ki-67 monoclonal antibody. Ki-67 is measured as a percentage of positive tumor cells. The investigator will conduct three paired t-tests comparing the percent Ki-67 at baseline to the percent Ki-67 after treatment. There will be one t-test for each arm.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Borges, MD, MSc, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Cancer Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No